CLINICAL TRIAL: NCT05435365
Title: An Observational Study Investigating The Experiences of Patients In Immunotherapy Clinical Trials
Brief Title: Investigating The Experiences of Patients In Immunotherapy Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 8328197
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Immunotherapy; Cancer
Keywords: Immunotherapy; Cancer; Diversity In Immunotherapy Clinical Trials
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has been observed before that participation in medical trials has been in favor of specific demographic groups. But research pointing out which trial attributes impact participation positively or negatively is sparse.

This study invites various participants to collect more data on their immunotherapy clinical experiences. The goal is to know which factors always limit how patients participate or complete the medical study they are first interested in.

The data obtained in the trial will be assessed through a variety of demographic lenses to discover patterns that might improve the experience of immunotherapy patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patient has self-identified as planning to participate in an interventional clinical trial using immunotherapy
* Patient has been diagnosed with a type of cancer
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient has an ECOG score of 4 or higher
* Patient is not able to provide consistent digital reporting as per study requirements
* Patient does not complete Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer who are actively considering enrolling in an immunotherapy interventional clinical trials, but have not yet completed enrollment and randomization in said clinical trial.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in an immunotherapy clinical trial | 3 months
Rate of patients who remain in immunotherapy clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loree JM, Anand S, Dasari A, Unger JM, Gothwal A, Ellis LM, Varadhachary G, Kopetz S, Overman MJ, Raghav K. Disparity of Race Reporting and Representation in Clinical Trials Leading to Cancer Drug Approvals From 2008 to 2018. JAMA Oncol. 2019 Oct 1;5(10):e191870. doi: 10.1001/jamaoncol.2019.1870. Epub 2019 Oct 10. PMID 31415071
- [Background] Hussain-Gambles M. Ethnic minority under-representation in clinical trials. Whose responsibility is it anyway? J Health Organ Manag. 2003;17(2):138-43. doi: 10.1108/14777260310476177. PMID 12916177
- [Background] Ma MA, Gutierrez DE, Frausto JM, Al-Delaimy WK. Minority Representation in Clinical Trials in the United States: Trends Over the Past 25 Years. Mayo Clin Proc. 2021 Jan;96(1):264-266. doi: 10.1016/j.mayocp.2020.10.027. No abstract available. PMID 33413830

DOCUMENTS (1):
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT05435365/ICF_000.pdf